CLINICAL TRIAL: NCT06146452
Title: Evaluation of Micronutrient Levels in Patients Hospitalized in the Pediatric Palliative Care Service.
Brief Title: Micronutrient Status in Pediatric Palliative Care
Status: Active, not recruiting | Type: Observational
Sponsor: Dr. Behcet Uz Children's Hospital (Other)
Responsible Party: Principal Investigator, Derşan Onur, Principal Investigator, Dr. Behcet Uz Children's Hospital
Other Study IDs: PPC Micronutrient
Record Dates: First submitted 2023-11-19; First posted 2023-11-24 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Palliative Care; Micronutrients; Pediatric
Keywords: Pediatric; Palliative Care; micronutriens
MeSH Terms: interventions — Nuclear Receptor Subfamily 4, Group A, Member 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric palliative care: pediatric palliative care patients hospitalized in the Pediatric Palliative Care Clinic
  Interventions: Other: Not

INTERVENTIONS:
Other: Not — Not

SUMMARY:
The goal of this observational study is to determine the micronutrient levels in patients in the Pediatric Palliative Care Clinic. The main question it aims to answer are:

• What is the frequency of micronutrient deficiencies in pediatric palliative care patients?

DETAILED DESCRIPTION:
Palliative care is an important health service provided with a multidisciplinary approach to improve the quality of life of children with progressive and life-threatening diseases and to manage symptoms effectively. This service aims to provide children with a good life experience by meeting the physical, psychological, social and spiritual needs of patients and their families.

Micronutrients contain important nutritional components such as vitamins, minerals and other nutrients that are essential for maintaining normal functions of the body. Micronutrient deficiencies affect at least half of children under five years of age. In a study conducted in pediatric oncology patients, micronutrient deficiency was shown to have a frequency of 74%, and selenium deficiency in particular negatively affected clinical outcomes. Contrary to recommended nutrient intakes (RNI) and expert opinion for healthy children, evidence-based recommendations for micronutrient requirements in critically ill children are not available. However, in pediatric palliative care, if the nutritional history indicates inadequate nutritional intake and/or growth indicates malnutrition, nutritional deficiencies that may have systemic effects, such as iron and vitamin B12 deficiency, need to be investigated.

This article aims to fill the gap in the literature by determining the micronutrient levels of pediatric palliative care patients hospitalized in the Pediatric Palliative Care Clinic. The research aims to contribute to a better understanding of the nutritional needs of patients in pediatric palliative care and to direct treatment approaches more effectively.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in a pediatric palliative care service

Exclusion Criteria:

* Patients who are hospitalized without having chronic, complex, progressive or life-threatening diseases (for off-label reasons)

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Our study will be carried out in the only pediatric palliative care center in Izmir that has been accepting patients since 2018. Our center is a clinic where palliative care patients (with chronic, complex, progressive or life-threatening diseases) between the ages of 1 month and 18 years who require hospitalization for various indications are managed with a multidisciplinary approach.
Sampling Method: Non-Probability Sample
Enrollment: 249 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
the presence of micronutrient deficiency | 12/01/2023-01/01/2024
  Presence of micronutrient deficiency in patients hospitalized in pediatric palliative care clinic

CONTACTS AND LOCATIONS:
Overall Officials: Derşan Onur, Principal Investigator — Dr. Behcet Uz Children's Hospital
Locations (1):
- Dr. Behcet Uz Children's Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Revuelta Iniesta R, Gerasimidis K, Paciarotti I, McKenzie JM, Brougham MF, Wilson DC. Micronutrient status influences clinical outcomes of paediatric cancer patients during treatment: A prospective cohort study. Clin Nutr. 2021 May;40(5):2923-2935. doi: 10.1016/j.clnu.2021.03.020. Epub 2021 Mar 20. PMID 33964502
- [Result] Marino LV, Valla FV, Beattie RM, Verbruggen SCAT. Micronutrient status during paediatric critical illness: A scoping review. Clin Nutr. 2020 Dec;39(12):3571-3593. doi: 10.1016/j.clnu.2020.04.015. Epub 2020 Apr 22. PMID 32371094
- [Result] Verbov J. More consultant dermatologists are needed. J R Coll Physicians Lond. 1990 Jul;24(3):249. No abstract available. PMID 2213683